CLINICAL TRIAL: NCT03196414
Title: Study of T Cells Targeting CD138/BCMA/CD19/More Antigens (CART-138/BCMA/19/More) for Chemotherapy Refractory and Relapsed Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: myeloma-01
Record Dates: First submitted 2016-10-19; First posted 2017-06-22 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2016-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CART-138/BCMA/19/more (Experimental)
  Interventions: Biological: CART-138/BCMA/19/more

INTERVENTIONS:
Biological: CART-138/BCMA/19/more — Cyclophosphamide，Fludarabine，CART-138/BCMA /19/more cells Cyclophosphamide: 300 mg/m2 IV over 30 minutes on days -5 , -4,and -3; Fludarabine: 30 mg/m2 IV over 30 minutes immediately following the cyclophosphamide on day -5, -4, and -3 Biological: Anti-CD138/BCMA/CD19/more total CART cells 5x106- 100x106 CAR+ T cells per kg of recipient bodyweight

SUMMARY:
Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells. Genetically engineered lymphocyte (CART) therapy has showed good safety and efficacy in treatment of lymphoma and acute lymphoblastic leukemia. Researchers want to see if this helps people with multiple myeloma.To test the safety and efficacy of giving targeting CD138 or B-cell maturation antigen or CD19 or more antigens T cells in treating patients with multiple myeloma that is refractory to further chemotherapy or relapsed(after stem cell transplantation or intensive chemotherapy).

DETAILED DESCRIPTION:
Adults ages 18-75 with Relapsed and/or Chemotherapy Refractory Multiple Myelomas.

Design:

Participants may be screened with:

Medical history Physical exam Blood and urine tests Heart tests Bone marrow sample Multiple scans and X-rays Lymphocytes are collected by apheresis from the enrolled patient or a healthy donor. Blood is removed through a needle in an arm. The rest of the blood is returned through a needle in the other arm.

The cells will be changed in a laboratory. Participants will get 2 chemotherapy drugs over 5 days. Two days later, participants will get an intravenous (IV) catheter in an arm. They will get the split doses CART cells on day0, day1, day2 through the IV in 1 infusion.

After this, participants will stay in the hospital for at least 9 days and stay nearby for 2 weeks. Then they will have blood tests and see a doctor.

Participants will visit the clinic at 1, 2, 3, 6, 9 and 12 months after the infusion, then every 6 months until two years after infusion. A bone marrow sample will be taken at the 3-month visit.

ELIGIBILITY:
Inclusion Criteria:

* CD138 or BCMA antigen positive multiple myeloma in patients with no available curative treatment options (such as autologous or allogeneic SCT).
* Relapsed and/or refractory multiple myeloma.
* Relapsed after prior autologous or allogenic SCT.
* Expected survival ≥ 3 months
* Creatinine < 2.0 mg/dl
* Blood coagulation function: PT and APTT < 2x normal
* Arterial blood oxygen saturation > 92%
* Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) < 3x normal
* Karnofsky scores ≥ 60 and ECOG score ≤ 2
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Patients should not take system chemotherapy in one month and immunotherapy in three months prior to CART cells infusion.
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* History of myocardial infarction and severe arrhythmia in half a year
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Patients with fever of unknown origin (T > 38℃)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine if there is grade 3 to 5 cytokine release syndrome | 2 weeks-12 months after initial dose
  Number of Patients With Grade 3 Through Grade 5 Cytokine Release Syndrome(CRS) That Are Related to Study Intervening Measures, Graded According to NCI CTCAE Version 4.0

SECONDARY OUTCOMES:
Investigators try to assess major reaction rate (MRR, PR+VGPR+CR) at the end of the research. | up to 24 weeks
  Number of Patients achieved major reaction rate (MRR;PR+VGPR+CR) According to IMWG response criteria at the end of the research.

OTHER OUTCOMES:
Investigators try to test CART 138 cells copies in vivo. | 2 years
  CART Cell survival time by testing CART-138/BCMA cells copies in vivo through PCR Method.

CONTACTS AND LOCATIONS:
Overall Officials: Fu cheng cheng, PhD, Principal Investigator — First Affiliated Hospital,Soochow University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Zhang C, Zhou J, Zhang J, Chen X, Chen J, Wang P, Sun X, Lou X, Qi W, Kang L, Yu L, Wu D, Li C. Case Report: Reversible Neurotoxicity and a Clinical Response Induced by BCMA-Directed Chimeric Antigen Receptor T Cells Against Multiple Myeloma With Central Nervous System Involvement. Front Immunol. 2021 Feb 25;12:552429. doi: 10.3389/fimmu.2021.552429. eCollection 2021. PMID 33717057